CLINICAL TRIAL: NCT06374082
Title: Efficacy of Instant Messaging Reinforcement on the Learning Outcomes of Smoking Cessation Counseling Training in Nursing Students: A Randomized Controlled Trial
Brief Title: Instant Messaging Reinforcement for Smoking Cessation Counseling Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HKWC-2024-179
Record Dates: First submitted 2024-04-11; First posted 2024-04-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation Counseling Ability; Smoking Cessation Counseling Practice
Keywords: instant messaging; nursing students; smoking cessation training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blinding technique will be used to conceal the allocation. Participants will not know which group they are in as placebo messages will be introduced. Using a central allocation web-based-controlled randomization, outcome assessors and data analysts will be blind to group allocation, only the principal investigator will be aware of who belongs to the control and intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): WhatsApp messages based on smoking cessation counseling Knowledge-Attitude-Practice (KAP)
  Interventions: Other: WhatsApp message
- Control group (Placebo Comparator): WhatsApp messages about generic mental health information
  Interventions: Other: WhatsApp message

INTERVENTIONS:
Other: WhatsApp message — Participants in the intervention group will receive 3 WhatsApp messages per week for six weeks after attending the standardized course training "Tobacco Dependency Nursing Intervention and Management (NURS8205)". These messages are about the core content of the course, including (1) Knowledge Themes: harmfulness of smoking and benefits of quitting, the fundamentals of nicotine addiction, smoking cessation counselling with the 5A model, and pharmacotherapy for smoking cessation; (2) Attitude Themes: nurses' role in smoking cessation and the importance of smoking cessation; and (3) Practice Themes: practical advice on counseling techniques, communication skills by motivational interviewing, local smoking cessation resources for referral.
  Participants in the control group will receive 3 WhatsApp messages about generic mental health information per week for six weeks after attending the standardized course training "Tobacco Dependency Nursing Intervention and Management (NURS8205)".

SUMMARY:
This research aims to assess the impact of instant messaging reinforcement on the learning outcomes of smoking cessation counseling (SCC) training among master of nursing (MN) students at the University of Hong Kong. The hypotheses suggest that this reinforcement can enhance students' SCC knowledge and techniques, improve their perception of SCC, and increase their application of SCC in clinical work.

The study is a pragmatic randomized controlled trial (RCT) with a 1:1 allocation ratio, using WhatsApp Messenger (WhatsApp) messages for intervention and control groups. The intervention group receives messages related to SCC, while the control group receives generic mental health information. The subjects are MN students enrolled in the "Tobacco Dependency Nursing Intervention and Management" course.

The study uses various tools for measurement, including Ecological momentary assessment (EMA) and Providers Smoking Cessation Training Evaluation (ProSCiTE). The main outcome measures include SCC practice frequency, SCC knowledge score, SCC attitude score, and SCC practice score.

Data analysis will be performed in Statistical Package for the Social Sciences (SPSS), using descriptive statistics, intention-to-treat analysis, Chi-square and t-tests, Cohen's d for effect size, and linear mixed models. The expected results suggest that instant messaging reinforcement will enhance SCC knowledge, attitude, and practice among MN students.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy of instant messaging reinforcement on the learning outcomes of smoking cessation counseling (SCC) training among master of nursing (MN) students at the University of Hong Kong.

Hypotheses to be tested: (1) Instant messaging reinforcement can increase MN students' mastery of SCC knowledge and techniques. (2) Instant messaging reinforcement can increase MN students' positive perception towards SCC and their willingness to provide SCC in their clinical work. (3) Instant messaging reinforcement can increase MN students' SCC practice, i.e. the frequency at which they perform Ask, Advise, Assess, Assist, and Arrange (5As), during their clinical work.

Design and subjects: This proposed study is a 2-arm, placebo-control, pragmatic randomized controlled trial (RCT) with a 1:1 allocation ratio. The intervention involves sending reinforcement WhatsApp messages to participants. To ensure that the subjects do not know their assigned group, the investigators also sent WhatsApp messages to the control group, but these messages are unrelated to smoking cessation counseling. The targeted subjects are MN students who are taking the course "Tobacco Dependency Nursing Intervention and Management (NURS8205)" in the spring semester of 2024. The course mentioned would be attended by all students regardless of their participation in this study.

Intervention group: 3 WhatsApp messages per week for six weeks after course training. These messages are about the core content of the course developed based on the Knowledge-Attitude-Practice (KAP) model.

Control group: WhatsApp messages about generic mental health information with the same frequency and schedule as the intervention group.

Instruments: Ecological momentary assessment (EMA) measurement of SCC practice frequency; Providers Smoking Cessation Training Evaluation (ProSCiTE); Self-compiled questionnaire on SCC knowledge; Self-compiled baseline questionnaire.

Main outcome measures: (1) MN students' SCC practice frequency, measured by EMA; (2) MN students' SCC knowledge score, measured by self-compiled questionnaire; (3) MN students' SCC attitude score, measured by attitude subscale of Providers Smoking Cessation Training Evaluation (ProSCiTE); (4) MN students' SCC practice score, measured by behavior subscale of Providers Smoking Cessation Training Evaluation (ProSCiTE).

Data analysis: Data analysis will be conducted in SPSS for Windows (version 20), using descriptive statistics (frequency, percentage, mean) to summarize outcomes and variables. Intention-to-treat analysis will handle participants lost to follow-up as no change. Outcome comparisons between groups will utilize Chi-square and t-tests, calculating Cohen's d for effect size. Linear mixed models will evaluate intervention effects on KAP, considering multiple observations and data clustering within subjects. SCC practice frequency, as measured by EMA, will be analyzed at between- and within-person levels using the "xtcenter" module, exploring associations with outcomes simultaneously.

Expected results: Instant messaging will improve MN students' SCC knowledge and skills, positive attitude toward providing SCC, and eventually increase their SCC practice frequency in their clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* MN students (1 or 2 years)
* Able to access WhatsApp and receive messages

Exclusion Criteria:

• Currently attending any other SCC training program other than this course

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-04-26 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
SCC practice measurement | The EMA will be conducted every night for two weeks after 6 weeks of instant messaging reinforcement
  Participants' SCC practice would be measured through ecological momentary assessment (EMA) by asking how many times they have performed Ask, Advise, Assess, Assist, and Arrange (5As) on each working day

SECONDARY OUTCOMES:
SCC knowledge score | through study completion, an average of 6 months
  Measured by self-compiled questionnaire on knowledge about SCC, the score ranges from 0 to 14, with higher score indicating better outcome
SCC attitude score | through study completion, an average of 6 months
  Measured by attitude subscale of Providers Smoking Cessation Training Evaluation (ProSCiTE), the score ranges from 8 to 40, with higher score indicating better outcome
SCC practice score | through study completion, an average of 6 months
  Measured by behavior subscale of Providers Smoking Cessation Training Evaluation (ProSCiTE), the score ranges from 19 to 95, with higher score indicating better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Derek Yee Tak CHEUNG, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong KongLKS Faculty of Medicine, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.
Access Criteria: Research data and documentation will be available upon request.